CLINICAL TRIAL: NCT02997956
Title: Phase IB/II Study of Tocilizumab in Patients With Hepatocellular Carcinoma (HCC) Undergoing Transarterial Chemoembolization (TACE)
Brief Title: Study of Tocilizumab in Patients With Hepatocellular Carcinoma (HCC) Undergoing Transarterial Chemoembolization (TACE)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding issues
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.105; HUM00104809 (Other: University of Michigan)
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Participants will receive Tocilizumab (ACTEMRA®) at 4, 6, or 8 mg/kg IV dose escalation on days 1, 29 and 57.
  The first part of the trial will be Phase Ib and will enroll 18 participants. Participants will receive TACE on day 1 and Tocilizumab at dose level 1, 2, or 3 on days 1, 29 and 57. Maximum tolerated dose (MTD) of Tocilizumab will be determined.
  The second part of the trial will be a Phase II and will enroll 50 subjects. Participants will receive TACE on day 1 and Tocilizumab at the MTD on days 1, 29 and 57.
  Interventions: Drug: Tocilizumab; Procedure: Transcatheter Arterial Chemoembolization

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive Tocilizumab (ACTEMRA®) at 4, 6, or 8 mg/kg IV dose escalation on days 1, 29 and 57.
  Other Names: ACTEMRA
Procedure: Transcatheter Arterial Chemoembolization — Minimally invasive procedure performed in interventional radiology to restrict a tumor's blood supply
  Other Names: TACE

SUMMARY:
This is a phase IB study design planned to identify the MTD (Maximum Tolerated Dose) of Tocilizumab in HCC (Hepatocellular Carcinoma) patients followed by a phase II design whereupon the primary objective will be median progression free survival (PFS).

DETAILED DESCRIPTION:
TACE (Transarterial Chemo Embolization) has shown to improve overall survival compared to non-treated patients with intermediate HCC (Hepatocellular Carcinoma) tumors. However, TACE is not considered a curative strategy and eventual local recurrence is observed in nearly all (>95%) of cases. Therefore, significant clinical equipoise exists in this large group of HCC patients such that novel therapies can be tested in an adjuvant manner to TACE. Based on pre-clinical data in HCC and the increasing identification that IL-6 signaling leads to tumor progression or local recurrence in other solid malignancies, significant rationale exists for the use of Tocilizumab, an IL-6 receptor inhibitor adjuvant to TACE. While Tocilizumab has been demonstrated to be safe in RA patients and is FDA approved, limited data exists for the maximum tolerated dose (MTD) in patients with cirrhosis and HCC. Therefore, a lead in phase IB study design is planned to identify the MTD of Tocilizumab in HCC patients followed by expansion to the phase II component whereupon the primary objective will be median progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of HCC, Barcelona-Clinic Liver Cancer (BCLC) stage B
* FFPE (Fixed-paraffin Embedded) tumor tissue (two cores preferred) for biomarker analysis
* Prior radioembolization, local ablative therapies (radiofrequency, microwave or cryoablation), radiation (external beam or stereotactic), or hepatic resection permitted if completed ≥ 4 weeks prior to study enrollment and if patient has recovered with ≤ grade 1 toxicity and if untreated measurable disease is present.
* Radiographically measurable disease by mRECIST in at least one site not previously treated by local therapies.
* Must not be receiving treatment with other investigational agents and must not have received any other investigational agent's ≤ 4 weeks prior to registration.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Required lab and acceptable range criteria.
* Women of child-bearing potential and men must agree to use 2 methods of adequate contraception.
* No contraindications to TACE therapy
* Child-Pugh Score A-B
* Ability to understand and the willingness to sign a written informed consent, and the willingness to comply with the requirements of the protocol.
* Life expectancy greater than 3 months.
* Adequate baseline organ and marrow function

Exclusion Criteria:

* History of hepatitis B
* Women must not be pregnant or breastfeeding
* Presence of other malignancies
* Active or history of Tuberculosis
* Patients with known HIV positive status
* Conditions with impaired immunity or on immunosuppressive medications such as oral steroids, calcineurin inhibitors, or anti-proliferative agents.
* Must have no evidence of significant, uncontrolled concomitant diseases
* Must have no ongoing or active, uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Tocilizumab | 84 Days Post Treatment
  The MTD is defined as the dose of Tocilizumab that induces dose-limiting toxicity in 20% of subjects or less when added to TACE. Patients must complete 84 days of treatment before the dose can be escalated.
Median Progression Free Survival | 2 Years Post Treatment
  Patients will be followed every 3 months for 2 years post treatment. Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death. Progressive disease is defined as at least a 20% increase in the sum of the LD or the appearance of one or more new lesions.

SECONDARY OUTCOMES:
Number of patients that respond to treatment | 2 Years Post Treatment
  Number of patients that respond to treatment
Number of patients alive at two years post treatment | 2 Years Post Treatment
  Number of patients alive at two years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Welling, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States